CLINICAL TRIAL: NCT02783859
Title: A Multi-centre Double-blind Randomised Controlled Trial to Determine if a Longer Duration of Amoxicillin-clavulanic Acid (Compared to Shorter Duration) Improves Clinical Outcomes of Children Hospitalised With Community-acquired Pneumonia
Brief Title: Hospitalised Pneumonia With Extended Treatment (HOPE) Study
Acronym: HOPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Griffith University (Other); Sarawak General Hospital (Other); University of Malaya (Other); The University of Queensland (Other); Queensland University of Technology (Other); Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HOPE_V5_01022017
Record Dates: First submitted 2016-05-05; First posted 2016-05-26 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia
Keywords: Children; Anti-Bacterial Agents; Indigenous Population; Hospitals
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active arm: Amoxicillin-clavulanic Acid (Experimental): 8 days of oral amoxicillin-clavulanic Acid 400/57 duo formulation (70-90mg/kg/day, twice daily dosing: max 980mg per day)
  Interventions: Drug: Amoxicillin-clavulanic Acid
- Placebo arm (Placebo Comparator): 8 days of oral placebo (equivalent volume as the active arm)
  Interventions: Drug: Placebo (for Amoxicillin-clavulanic Acid)

INTERVENTIONS:
Drug: Amoxicillin-clavulanic Acid
  Arms: Active arm: Amoxicillin-clavulanic Acid
Drug: Placebo (for Amoxicillin-clavulanic Acid)
  Arms: Placebo arm

SUMMARY:
An intervention study to determine if a longer duration of antibiotics (compared to shorter duration) improves the short and long term clinical outcomes of children hospitalised for pneumonia

DETAILED DESCRIPTION:
A multi-centre double-blind randomised controlled trial to determine if a longer duration of amoxicillin-clavulanic acid (compared to shorter duration) improves the short and long term clinical outcomes of children hospitalised with community-acquired pneumonia, in Indigenous children and a developing country

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalised children aged 3-mo to 5-yrs (in Darwin, children have to be Indigenous)
2. Have features of severe pneumonia on admission (temperature >37.5 celsius or a history of fever at home or observed at the referring clinic, age-adjusted tachypnoea [respiratory rate>50 if <12-months; respiratory rate>40 if >12-months] with chest wall recession and/or oxygen saturation <92% in air), and consolidation on chest X-ray as diagnosed by treating clinician
3. After 1-3 days of IV antibiotics, are afebrile, with improved respiratory symptoms and signs, oxygen saturation>90% in air and are ready to be switched to oral amoxicillin-clavulanate, and
4. Have symptoms of no longer than 7 days at point of hospitalisation.

Exclusion Criteria:

1. Current wheeze
2. Underlying chronic illness other than asthma (e.g. bronchiectasis, cyanotic congenital heart disease or cardiac failure, neuromuscular disorders, immunodeficiency) that could potentially influence the current illness
3. Severe malnutrition (weight-for-height Z-score <-3)
4. Complicated (effusion, empyema or abscess) pneumonia, including tuberculosis
5. Extra-pulmonary infection requiring antibiotic therapy (e.g. meningitis)
6. Beta-lactam allergy
7. Previously enrolled
8. Lack a mobile phone and/or unable to return for follow-up clinic visits during the next 24 months

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
The proportion without chronic respiratory symptoms and signs or bronchiectasis. | Clinical review at 24 months (range 23-25 months)
  Any further chronic respiratory symptoms and signs or bronchiectasis though the child's medical records (community or hospital) will be captured. These children will be reviewed at 24 months, however many children will reside in geographically isolated locations, thus a range of 23-25 months is a reasonable timeframe to capture clinically important outcomes.

SECONDARY OUTCOMES:
The proportion with clinical cure (i.e. complete resolution of respiratory symptoms and signs). | Clinical review week 4 (range 4-6 weeks)
  Children will have a standardised respiratory clinical assessment, completed by either a member of the study team or health provider. These children will be reviewed at week 4, however many children will reside in geographically isolated locations, thus a range of 4-6 weeks is a reasonable time frame to capture clinically important outcomes.
Time to next respiratory-related hospitalisation assessed by chart reviews | Clinical review week 4 (range 4-6 weeks)
  Data will be captured through chart reviews of children's medical records (e.g. hospital and/or community health record) and/or information from parents in next 12 months
Adverse events | Adverse events monitored while participant taking trial medication
  Adverse effects will be monitored (anorexia, nausea, vomiting, abdominal pain, diarrhoea, rashes) while children are actively taking trial medication (e.g. 8 days). Parents will also keep a diary of adverse events.
Nasopharyngeal bacteria antibiotic resistance patterns | Baseline (admission to hospital, week 4 (range 4-6 weeks) and 12 months (range 12-14 months)
  Nasopharyngeal respiratory antibiotic resistance will be assessed using nasal swabs. Nasopharyngeal respiratory bacterial pathogens and antibiotic resistance will be assessed using research laboratory's previously published methods.
Gene expression data | Baseline (hospital admission) and 4-6 weeks (where possible)
  Gene expression micro-arrays will be performed in a subgroup of children (where bloods can be obtained)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chang, PhD, Principal Investigator — Menzies School of Health Research
Locations (5):
- Menzies School of Health Research, Darwin, Northern Territory, Australia
- Malaysia (3):
  - University Malaya Medical Centre and Klang Hospital, Kuala Lumpur, Kuala Lumpur
  - Sabah Women and Children's Hospital, Kota Kinabalu, Sabah
  - Sarawak General Hospital, Sibu, Sarawak
- Starship Children's Hospital & KidzFirst Hospital, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No